CLINICAL TRIAL: NCT01265654
Title: Reasons for Changing HOrmonal Therapy of Advanced Breast Cancer
Acronym: HOT ABC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCZ-FAS-2010/1
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer; Hormonal Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- All patients: Patients with ABC and two lines of hormonal treatment

SUMMARY:
Breast cancer is the leading type of cancer in women. Although big advance in diagnostics and treatment of early and breast cancer has been made in recent years breast cancer still has a significant mortality rate. A number of treatment modalities exist for postmenopausal women with advanced breast cancer. The treatment modality is chosen based on patient and tumour characteristics. Hormonal treatment is preferred and recommended in women with hormone sensitive breast cancer (ESMO, CECOG and NCCN guidelines). Tumor markers are an established method of monitoring systemic therapies in various cancers. Tumor markers CA 15-3 and CEA are used in clinical practice to monitor treatment efficacy of metastatic breast cancer. Blood levels of tumor markers are widely used to assess response/progression to treatment and guide therapy change. Treatment efficacy is assessed by imaging methods in clinical studies. Change of therapy in clinical study is usually done when progression based on RECIST criteria is found. Hormonal treatment has slower onset of effect compared with chemotherapy that can last several weeks. Also when a new therapy is started spurious early rises may occur. Therefore rising levels of tumor markers during the first weeks of new hormonal therapy are not necessarily sign of progression and should not be the only guidance for treatment change. Evidence of treatment efficacy form clinical studies and treatment change is based on imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least two finished lines of hormonal treatment for advanced breast cancer Tumor markers (CEA. CA15-3) values available at the time of onset and discontinuation of therapy Imaging methods results available at the time of onset and discontinuation of therapy

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with hormone sensitive advanced breast cancer that have been treated with minimum two hormonal agents according to approved SmPC.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Reasons for change of hormonal therapy (biochemical progression, objective progression, symptomatic progression, safety reasons, other) | Every 3 months

SECONDARY OUTCOMES:
Changes in values of tumor markers (CEA, CA 15.3) | Every 3 months.
Time to progression | Every 3 months
Type of hormonal treatment | Every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ales Kminek, Study Director — AstraZeneca Czech Republic; Katarina Petrakova, Principal Investigator — Masaryk Memorial Cancer Institute, Brno, Czech Rep.; Lubos Petruzelka, Principal Investigator — General Teaching Hospital, Prague, Czech Rep.
Locations (37):
- Czechia (37):
  - Research Site, Benesov U Prahy
  - Research Site, Brno
  - Research Site, Cheb
  - Research Site, Chomutov
  - Research Site, České Budějovice
  - Research Site, Český Krumlov
  - Research Site, Fryštát
  - Research Site, Havlíčkův Brod
  - Research Site, Hradec Králové
  - Research Site, Jablonec nad Nisou
  - Research Site, Jičín
  - Research Site, Jihlava
  - Research Site, Kladno
  - Research Site, Kolín
  - Research Site, Liberec
  - Research Site, Most
  - Research Site, Náchod
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Opava
  - Research Site, Ostrava
  - Research Site, Ostrava - Fifejdy
  - Research Site, Ostrava - Vitkovice
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Písek
  - Research Site, Prague
  - Research Site, Prostějov
  - Research Site, Přerov
  - Research Site, Rakovník
  - Research Site, Sokolov
  - Research Site, Strakonice
  - Research Site, Šumperk
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
  - Research Site, Zlín
  - Research Site, Znojmo